CLINICAL TRIAL: NCT02895711
Title: Radiation Doses of Pediatric Patients During Ureteroscopy and Percutaneous Nephrolithotomy
Brief Title: Radiation Dose of Pediatric Patients During Ureteroscopy
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Rajeev Chaudhry, Assistant Professor, University of Pittsburgh
Other Study IDs: PRO10040374
Record Dates: First submitted 2016-08-30; First posted 2016-09-12 (Estimated); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with urolithiasis: To record the effective radiation dose to the patient during endourologic procedures to treat urolithiasis

SUMMARY:
The purpose of this study is to quantify the radiation exposure from diagnostic testing and surgical treatment during routine endourologic procedures for symptomatic urolithiasis.

DETAILED DESCRIPTION:
Routine endourologic procedures will be performed at the Childrens Hospital of Pittsburgh by one of the investigators listed on this study. Fluoroscopic radiation exposure during these procedures is used to guide the surgical devices that are used to treat the stones. The investigators will be measuring the radiation effective skin dose by two methods. First, the investigators will place two "Microdot" thermal leak detectors (TLD) on the patient. These devices which are the size and thickness of a dime will be within plastic bags taped to the patients body within the central focus of the fluoroscopy image. At the completion of the procedure the TLD's will be transferred to the Radiation Safety Office in Oakland to be read and the dose recorded.

Second, a flat chamber that is integral with all fluoroscopy machines used at Children's Hospital will measure the dose-area product (DAP) for each case which will allow us to calculate the effective dose. This device is a component of the colimeter on the arm of the x-ray machine used for fluoroscopy. It measures the radiation that is returned to the x-ray machine and calculates the dose delivered to the patient by comparing the amount delivered to the patient to the amount returned to the machine. Its use is automatic when any x-rays are delivered and does not involve any manipulation of the patient or alteration of normal procedure.

No additional procedures or change in duration is necessary for this study

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects will be male and female volunteers of 0-18 years of age with documented urolithiasis who is undergoing a urologic procedure that utilizes fluoroscopy radiation.
* The racial, gender and ethnic characteristics of the proposed subject population reflect the demographics of Pittsburgh and the surrounding area and/or the population of the University of Pittsburgh.
* We shall attempt to recruit subjects in respective proportion to these demographics.

Exclusion Criteria:

* None

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with urolithiasis
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2010-09; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Exposed to fluoroscopic radiation | through study completion, an average of 1 year
  To record the effective radiation dose to the patient during endourologic procedures to treat urolithiasis

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Chaudhry, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No